CLINICAL TRIAL: NCT05699460
Title: A Pre-Gene Therapy Study of Early Parkinson's or Multiple System Atrophy Progression by Longitudinal Clinical and Biomarker Assessments
Brief Title: Pre-Gene Therapy Study in Parkinson's Disease and Multiple System Atrophy
Status: Active, not recruiting | Type: Observational
Sponsor: AskBio Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: ASK-PD-0-CS-001
Record Dates: First submitted 2022-10-13; First posted 2023-01-26 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Parkinson's Disease; Multiple System Atrophy, Parkinson Variant; Multiple System Atrophy
Keywords: MSA; MSA-P; PD; Observational; Natural History
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early Parkinson's disease
  Interventions: Other: This is an observational study.
- Possible or Probable MSA-P
  Interventions: Other: This is an observational study.

INTERVENTIONS:
Other: This is an observational study. — This is an observational study.

SUMMARY:
The objective of this study is to describe disease progression in study participants diagnosed with early Parkinson's Disease or Multiple System Atrophy - Parkinsonian Type up to 18 months as delineated by clinical and biochemical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Idiopathic PD
* Diagnosis of MSA-P
* One to six years from clinical diagnosis of PD
* Less than 4 years from clinical diagnosis of MSA with expected survival >3 years
* Stable medication regimen
* Ability to walk with or without an assistive device

Exclusion Criteria:

* Movement disorder due to known cerebrovascular disease, brain tumor, trauma, exposure to parkinsonian-linked toxicants or other neurological diseases
* Presence of dementia, psychosis, substance abuse or poorly controlled depression
* Prior brain surgery (i.e. deep brain stimulation) or other brain imaging abnormalities
* History of cancer or poorly controlled medical conditions
* Receiving an investigational drug

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will have a diagnosis of early Parkinson's disease OR possible or probably MSA-P
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Motor symptoms as assessed by the Movement Disorder Society's Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | 18 months
  Change from baseline in the MDS-UPDRS. The MDS-UPDRS contains 4 subscales: Part I, non-motor aspects of experiences of daily living (13 items); Part II, motor aspects of experiences of daily living (13 items); Part III, motor examination (33 scores based on 18 items); Part IV, motor complications (6 items). The rating for each item, or sub-item, is from 0 (normal) to 4 (severe). The total score for each Part is obtained from the sum of the corresponding item scores.
MSA symptoms/signs as assessed by the Unified Multiple System Atrophy Rating Scale (UMSARS) | 18 Months
  Change from baseline in the Unified Multiple System Atrophy Rating Scale (UMSARS) and compared to placebo. UMSARS total scores range from 0-104 points with higher scores indicating greater severity of impairment.

SECONDARY OUTCOMES:
Change in the quality of life as measured by Parkinson's Disease Questionnaire (PDQ-39) | 18 months
  Change from baseline in the Parkinson's Disease Questionnaire (PDQ-39). PDQ-39 is a self-reported 39-item questionnaire designed to measure health related quality of life in Parkinson's Disease patients. It provides scores in 8 domains: mobility, activities of daily living, emotions, stigma, social support, cognitive function, bodily discomfort and communication, as well as a summary index score for quality of life.
Change in the quality of life as measured by Multiple System Atrophy Quality of Life (MSA-QoL) | 18 months
  Change from baseline in the Multiple System Atrophy Quality of Life (MSA-QoL) scale. MSA-QoL is a self-reported questionnaire that measures MSA impact in day to day activities. Scale consists of 40 items with a five response option format (0 - no problem to 4 extreme problem) and a "not applicable" response option.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (7):
  - University of California Irvine, Irvine, California
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Quest Research Institute, Farmington Hills, Michigan
  - Ohio Health Research Institute, Columbus, Ohio
  - OHSU Parkinson Center & Movement Disorders Program, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Poland (4):
  - Zespol Poradni Specjalistycznych - Botaniczna 3 Poradnia Neurologiczna Szpital Uniwersytecki w Krakowie, Krakow, Lesser Poland Voivodeship
  - Specjalistyczna Praktyka Lekarska, Prof. Grzegorz Opala, Katowice
  - Mazowiecki Szpital Bródnowski w Warszawie, Oddział Neurologii, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny im. prof. Witolda Orłowskiego, Oddział Neurologii i Epileptologii, Warsaw

IPD SHARING:
Plan to Share IPD: No